CLINICAL TRIAL: NCT00662935
Title: Evaluation of Efficacity and Safety of Deep Brain Stimulation (DBS) in Chronic and Treatment-Resistant Cluster Headache(CH)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Collaborators: Medtronic (Industry)
Responsible Party: GIRAN Cynthia, Département de la Recherche Clinique et de l'Innovation
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 04 -APN -03
Record Dates: First submitted 2008-04-17; First posted 2008-04-21 (Estimated); Last update posted 2008-04-21 (Estimated); Status verified 2008-04

CONDITIONS: Cluster Headache
Keywords: deep brain stimulation; cluster headache; hypothalamus
MeSH Terms: conditions — Cluster Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Experimental): the sequence of stimulation begins by OFF
  Interventions: Procedure: setting-up of an electrode in deep brain
- 1 (Experimental): the sequence of stimulation begins by ON
  Interventions: Procedure: setting-up of an electrode in deep brain

INTERVENTIONS:
Procedure: setting-up of an electrode in deep brain — deep brain stimulation of the postero-inferoir hypothalamus

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of deep brain stimulation (DBS) in chronic and treatment-resistant CH. Inclusion criteria are: patients with chronic CH (>3years), with daily attack and non response to adequate treatment. Electrodes are implanted stereotactically in the postero-inferior hypothalamus. In this crossover, randomized, placebo-controlled double-blinded study, the efficacy of DBS is evaluated using comparison of two one-month sequences: one with stimulation "on" and the other with stimulation "off" (placebo sequence). Efficacy is defined as ≥50% decrease of weekly frequency of CH attacks. After the randomized period, long-term efficacy and safety are evaluated after one year of stimulation in open conditions.

DETAILED DESCRIPTION:
Over the past 7 years, deep brain stimulation (DBS) has been used in various centres to treat patients with intractable chronic cluster headache (CH). Results in these non-controlled studies were encouraging but need to be confirmed in controlled conditions. The aim of this study is to evaluate the efficacy and safety of DBS in chronic and treatment-resistant CH, in randomized placebo-controlled conditions.

Inclusion criteria are: patients with chronic CH (>3years), with daily attack and non response to adequate treatment (verapamil up 960 mg/d, lithium with plasmatic level 0.6-1 mEq/ ml, and association of both drugs). After induction of local anaesthesia, electrodes are implanted stereotactically in the postero-inferior hypothalamus according to the previously described coordinates, and connected to a sub-cutaneous generator. In this crossover, randomized, placebo-controlled double-blinded study, the efficacy of DBS is evaluated using comparison of two one-month sequences: one with stimulation "on" and the other with stimulation "off" (considered as the placebo sequence). Primary efficacy is defined as ≥50% decrease of weekly frequency of CH attacks, compared to a prospective run-in pre-implantation period. Safety and tolerability are clinically and biologically assessed. After the randomized period, long-term efficacy and safety are evaluated after one year of stimulation in open conditions.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 65 year old
* suffering from cluster headache since 3 years at least
* not responding to others treatments such as : verapamil, lithium or both of them

Exclusion Criteria:

* patient with addiction
* pregnancy or feeding women
* contraindication to general anesthetic
* contraindication to MRI

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-05; Primary Completion 2008-01 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Decrease (≥50% by reference to a prospective pre-implantation run-in period) of the weekly frequency of cluster headache attacks between treatment and placebo one-month sequences. | between treatment and placebo one-month sequences.

SECONDARY OUTCOMES:
Intensity of dysautomic dysfunction, acute treatment consumption, quality of life Between treatment and placebo one-month sequences. | Between treatment and placebo one-month sequences.

CONTACTS AND LOCATIONS:
Overall Officials: Michel LANTERI-MINET, PhD, Principal Investigator — Department of Neurology, CHU de NIce; Denys FONTAINE, PhD, Principal Investigator — Department of Neurology, CHU de Nice

REFERENCES:
- [Derived] Fontaine D, Lazorthes Y, Mertens P, Blond S, Geraud G, Fabre N, Navez M, Lucas C, Dubois F, Gonfrier S, Paquis P, Lanteri-Minet M. Safety and efficacy of deep brain stimulation in refractory cluster headache: a randomized placebo-controlled double-blind trial followed by a 1-year open extension. J Headache Pain. 2010 Feb;11(1):23-31. doi: 10.1007/s10194-009-0169-4. PMID 19936616